CLINICAL TRIAL: NCT06444763
Title: Effect of Maolactin™ FMR Supplementation on Exercise Recovery, Inflammation, and Muscle Comfort in an Otherwise Healthy Population: A Double-blind Randomized Placebo-controlled Study
Brief Title: Effect of Maolactin™ FMR on Exercise Recovery, Inflammation and Muscle Comfort in an Otherwise Healthy Population
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAOJOI(B)
Record Dates: First submitted 2024-05-24; First posted 2024-06-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: Chronic Inflammation; Mobility; Muscle Pain; Joint Pain
MeSH Terms: conditions — Myalgia; Arthralgia | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maolactin (Experimental): 2 capsules containing a total of 500 mg/day active proteins taken once daily before the morning meal
  Interventions: Drug: Maolactin
- Maltodextrin (Placebo Comparator): 2 capsules containing maltodextrin (0mg/day active proteins) taken once daily before the morning meal
  Interventions: Drug: Maltodextrin

INTERVENTIONS:
Drug: Maolactin — Once daily dose of 2 capsules containing a total of 500mg/day Maolactin
  Arms: Maolactin
Drug: Maltodextrin — Once daily dose of 2 capsules of Maltodextrin containing a total of 0mg/day Maolactin
  Arms: Maltodextrin

SUMMARY:
This is a double blind, randomised, placebo-controlled, parallel-group trial to evaluate the effect of Maolactin FMR supplementation on chronic inflammation, mobility and muscle and joint pain in an otherwise healthy population of adults over 45 years old over 10 weeks with 8 weeks supplementation.

This is PART B of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 45 years and older
* Generally healthy
* BMI 25.0 - 35.0 kg/m2
* C-reactive protein (CRP) equal to or greater than 2.0 mg/L
* Feel pain or discomfort in joints/muscle for at least 3 months
* Able to provide informed consent
* Agree not to change current diet and/or exercise frequency or intensity during study period
* Agree to not participate in another clinical trial while enrolled in this trial

Exclusion Criteria:

* Serious illness(1) e.g., mood disorders such as depression, anxiety or bipolar disorder, neurological disorders such as MS, kidney disease, liver disease or heart conditions
* Unstable illness(2) e.g., diabetes and thyroid gland dysfunction
* Unstable intake of any medication or supplement(3)
* Acute injuries on reporting area
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy including low dose aspirin
* Receiving medications known to affect inflammation such as steroids
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>21 alcoholic drinks per week)
* Pregnant or lactating women
* Allergic to any of the ingredients in active or placebo formula
* Participants who are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 1 month
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion

  1. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.
  2. An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity.
  3. An unstable intake is any dose that has changed by more than 10% of the previous dose in the past 4-weeks

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Inflammatory status | Baseline and Week 8
  Change in Inflammatory status as assessed by C-reactive protein (CRP) via blood test

SECONDARY OUTCOMES:
Change in Weight | Baseline and Week 8
  Change in Weight as measured by digital scales
Change in Body Mass Index (BMI) | Baseline and Week 8
  Change in BMI as assessed by digital scale for weight and stadiometer for height
Change in Musculoskeletal Health Questionnaire (MSK-HQ) | Baseline, Week 4 and Week 8
  Change in MSK-HQ as self-reported by participants. Scored on a range of 0-56, with a higher score indicating health status.
Change in Visual Analogue Scale (VAS) Muscle Pain | Baseline, Week 4 and Week 8
  Change in VAS Muscle Pain as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of muscle pain.
Change in Visual Analogue Scale (VAS) Pain | Baseline, Week 4 and Week 8
  Change in VAS Pain as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of pain
Change in Visual Analogue Scale (VAS) Fatigue | Baseline, Week 4 and Week 8
  Change in VAS Fatigue as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of fatigue.
Change in Visual Analogue Scale (VAS) Mobility | Baseline, Week 4 and Week 8
  Change in VAS Mobility as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of mobility.
Change in Visual Analogue Scale (VAS) Stiffness | Baseline, Week 4 and Week 8
  Change in VAS Stiffness as self-reported by participants. Minimum score = 0, Maximum score = 10. Higher scores indicate a higher level of stiffness.
Change in Multidimensional Fatigue Inventory (MFI) | Baseline, Week 4 and Week 8
  Change in MFI as self-reported by participants. Comprises 20 questions rated on a 5 point scale. with a higher score indicating a higher level of fatigue.
Change in Blood Pressure (BP) | Baseline and Week 8
  Change in BP as assessed by digital blood pressure monitor
Change in Heart Rate (HR) | Baseline and Week 8
  Change in HR as assessed by digital heart rate monitor
Change in Oxygen Saturation | Baseline and Week 8
  Change in Oxygen Saturation as measured by pulse oximeter
Change in Cytokines | Baseline and Week 8
  Change in Cytokines as measured by blood test
Change in Monocyte Chemotactic Protein-1 (MCP-1) | Baseline and Week 8
  Change in MCP-1 as measured by blood test
Change in Nuclear Factor KappaB (NF-kB) | Baseline and Week 8
  Change in NF-kB as measured by blood test
Change in P-selectin | Baseline and Week 8
  Change in P-selectin as measured by blood test
Change in E-selectin | Baseline and Week 8
  Change in E-selectin as measured by blood test
Change in Matrix Metalloproteinase-3 (MMP3) | Baseline and Week 8
  Change in MMP3 as measured by blood test
Change in Cartilage Oligomeric Matrix Protein (COMP/thrombospondin-5) | Baseline and Week 8
  Change in COMP as measured by blood test
Change in Type II procollagen (CPII) | Baseline and Week 8
  Change in CPII as measured by blood test
Change in Type II collagen (C2C) | Baseline and Week 8
  Change in C2C as measured by blood test
Change in Creatine Kinase (CK) | Baseline and Week 8
  Change in CK as measured by blood test
Change in Myoglobin | Baseline and Week 8
  Change in Myoglobin as measured by blood test
Change in Full Blood Count (FBC) | Baseline and Week 8
  Change in FBC as measured by blood test
Change in Platelet agglomeration | Baseline and Week 8
  Change in Platelet agglomeration as measured by blood test
Change in Lipoprotein-associated phospholipase A2 (Lp-PLA2) | Baseline and Week 8
  Change in Lp-PLA2 as measured by blood test
Change in Intercellular Cell Adhesion Molecule-1 (ICAM-1) | Baseline and Week 8
  Change in ICAM-1 as measured by blood test
Change in Intercellular Cell Adhesion Molecule-2 (ICAM-2) | Baseline and Week 8
  Change in ICAM-2 as measured by blood test
Change in Vascular Cell Adhesion Molecule-1 (VCAM-1) | Baseline and Week 8
  Change in VCAM-1 as measured by blood test
Change in Vascular Cell Adhesion Molecule-2 (VCAM-2) | Baseline and Week 8
  Change in VCAM-2 as measured by blood test
Change in Platelet Endothelial Cell Adhesion Molecule-1 (PECAM-1) | Baseline and Week 8
  Change in PECAM-1 as measured by blood test
Change in Erythrocyte Sedimentation Rate (ESR) | Baseline and Week 8
  Change in ESR as measured by blood test
Change in Lactate Dehydrogenase (LDH) | Baseline and Week 8
  Change in LDH as measured by blood test
Change in P38 Mitogen-activated Protein Kinases (P38) | Baseline and Week 8
  Change in P38 as measured by blood test
Change in Electrolytes and Liver Function Tests (E/LFT) | Baseline and Week 8
  Change in E/LFT as measured by blood test
Change in 2 minute walk test | Baseline and Week 8
  Change in 2 minute walk test as measured by exercise testing
Change in sit-to-stand test | Baseline and Week 8
  Change in sit-to-stand test as measured by exercise testing
Change in Hand Grip Strength | Baseline and Week 8
  Change in Hand Grip Strength as measured by dynamometer
Change in Adverse Events | Baseline to week 8
  Change in Adverse Events self-reported by participants
Change in Gastrointestinal Tolerance | 1 week after starting product and Week 8
  Change in Gastrointestinal Tolerance as measured by Gastrointestinal Tolerance (GIT) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Briskey, PhD, Principal Investigator — RDC Clinical Pty Ltd
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia